CLINICAL TRIAL: NCT00452478
Title: A Phase IV, Open-Label, Multi-Centre Trial Evaluating the Conversion From Standard Phosphate Binder Therapy to Fosrenol® in Chronic Kidney Disease Stage 5 Patients on Haemodialysis
Brief Title: Conversion From Standard Phosphate Binder Therapy to Fosrenol® (Lanthanum Carbonate) in Chronic Kidney Disease Stage 5
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was stopped by the sponsor based on a non-safety related corporate decision
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-403; 2006-003364-64 (EudraCT Number)
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Kidney Diseases
Keywords: Hyperphosphataemia
MeSH Terms: conditions — Kidney Diseases; Hyperphosphatemia | interventions — lanthanum carbonate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate — 2250mg/day starting dose of lanthanum carbonate administered orally, in divided doses, with meals (500mg 750mg and 1000mg strengths)for 2 weeks; dose titration will occur based on serum phosphorus results not to exceed 3000mg/day.
  Other Names: FOSRENOL

SUMMARY:
The main aim of this research study is to see if giving Fosrenol®, a chewable tablet, to patients on haemodialysis works as well as other treatments currently used to lower blood phosphorus levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects greater than or equal to 18 years of age receiving a stable regimen of haemodialysis for chronic kidney disease (CKD) Stage 5 (defined as haemodialysis two or three times per week for at least two months prior to screening).
* Females of child bearing potential (FOCP) must be non-pregnant, non-lactating, have a negative serum beta human chorionic gonadotropin (HCG) test, and agree to comply with any applicable contraceptive requirements of the protocol.
* Subjects on a stable phosphate binder dose (defined as no change in medication or dosage for at least the one month prior to screening) with a serum phosphorus level between greater than 1.78 and less than or equal to 2.43 mmol/L (5.5 and 7.5 mg/dL).

Exclusion Criteria:

* Subjects with a corrected serum calcium level less than 2.1 mmol/L (8.5 mg/dL).
* Subjects with an intact parathyroid hormone (iPTH) level greater than 500 pg/mL, or a history of previous parathyroidectomy within 12 months of screening.
* Subjects with any significant bowel obstruction, active inflammatory bowel disease, gastrointestinal (GI) motility disorders, abnormal or irregular bowel motion, or a history of major GI surgery within the last 6 months will be excluded.
* Subjects receiving aluminium, magnesium, or combination therapy other than sevelamer hydrogen chloride (HCl) and calcium as a phosphate binder at the time of screening will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-05-22 (Actual); Primary Completion 2007-12-10 (Actual); Study Completion 2007-12-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving serum phosphorus levels of less than or equal to 1.78 mmol/L (5.5 mg/dL) following treatment with Fosrenol at Week 12 compared to treatment with their previous phosphate binder therapy | 12 weeks

SECONDARY OUTCOMES:
The maintenance of mean serum phosphorus levels following treatment with 2250 mg/day of Fosrenol | at Week 2 compared to baseline
Biochemical and haematological parameters | measured throughout the study
Assess safety & tolerability | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- Austria (2):
  - Landeskrankenhaus Feldkirch, Abteilung fur Nephrologie und dialyse, Feldkirch Tisis
  - Krankenhaus Elisabethinen/Dialysestation, Linz
- Ziekenhuis Zuid Oost Limburg, Genk, Belgium
- Denmark (3):
  - Frederica Sygehus, Fredericia
  - Holbaek Sykehus, Holbæk
  - Sygehus Viborg, Viborg
- Germany (6):
  - Dialysezentrum Barmbek, Hamburg
  - Dialysezentrum Heilbronn, Heilbronn
  - Dialyse Leipzig, Leipzig
  - Nephrologisches Zentrum Emsland, Lingen
  - nephrologische Schwerpunktpraxis, Oldenburg
  - diabetologische Schwerpunktpraxis, Villingen-Schwenningen
- University of Milan, San Paolo Hospital, Renal Division, Milan, Italy
- Gelre Ziekenhuizen, Apeldoorn, Netherlands